CLINICAL TRIAL: NCT05485129
Title: Use of HRV Measuring Hearing-aid Device to Detect Acute Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, Professor, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SQUID
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: BIORICS

INTERVENTIONS:
Device: BIORICS — Wearing BIORICS in their ear and perform mental arrhythmic test, relaxation exercises and Stroop test

SUMMARY:
Validation of in-ear device to measure acute mental stress in comparison with a Polar H10 chest band. Stress is measured on the basis of heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Dutch speaking and understanding
* Evidence of a personally signed and dated informed consent, indicating that the subject (or a legally recognized representative) has been informed of all pertinent aspects of the study
* Age ≥ 50 years
* No contra-indications for the use of the receiver in-the-ear device (BiometRIC SR 26UAA01GF), and smartwatch and chest strap heartrate monitor

Exclusion Criteria:

* • Smokers

  * Obese patients (BMI >30 kg/m2)
  * Presence of a pacemaker
  * Supraventricular tachycardias: atrial fibrillation, atrial flutter, frequent supraventricular extrasystole or frequent ventricular extrasystole
  * Otologic contraindications determined by licensed otolaryngologist

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability measured BIOMETRIC in-ear device | 1 day
  RMSSD

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No